CLINICAL TRIAL: NCT01833416
Title: Natural History of Cytomegalovirus (CMV) Infection and Disease Among Renal Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Helio Tedesco Silva Junior (Other)
Responsible Party: Sponsor-Investigator, Helio Tedesco Silva Junior, PhD, Hospital do Rim e Hipertensão
Organization: Hospital do Rim e Hipertensão (Other)
Other Study IDs: 2013027692
Record Dates: First submitted 2013-03-07; First posted 2013-04-16 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Infection in Solid Organ Transplant Recipients
Keywords: CMV infection; CMV disease; Natural history; Kidney transplant
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Although the accumulated knowledge regarding Cytomegalovirus (CMV) infection increased substantially over the past years, several issues still deserve further investigation. The epidemiology of this disease has been changing, perhaps influenced by new immunosuppressive strategies currently used and growing and widespread use of prophylaxis. The knowledge of the CMV viral load kinetics, using a polymerase chain reaction (PCR-based assay), among renal transplant recipients not receiving any prophylactic therapy will allow the determination of risk factors for and the impact of earlier intervention on CMV infection and disease. The goal is to ultimately improve the clinical outcomes for renal transplant recipients.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) infection remains one of the most common complications affecting organ transplant recipients, with significant morbidity and occasional mortality. The adverse impact of CMV infection on graft function underscores the importance of CMV on transplant outcomes.

CMV prevention strategies have resulted in significant reductions in CMV disease and CMV-related mortality. The reduction in the incidence of "indirect effects" of CMV infection has also been attributed to the use of CMV prevention. Nevertheless, management of CMV infection varies considerably among transplant centers. Two major strategies are commonly used for prevention of CMV: universal prophylaxis and preemptive therapy. Within each of these strategies, significant variation in clinical practice exists, including type of cellular or molecular diagnostics, antiviral therapies, monitoring and criteria for stopping treatment.

Although the use of universal prophylaxis has increased since the availability of valganciclovir, there is still a debate regarding the superiority of this strategy over the preemptive approach. Furthermore, this costly therapy or any other CMV prophylaxis is currently not reimbursed by our unified public health system. Therefore our strategy has been to use preemptive therapy. Additionally, because we consider different immunosuppressive regimens according to pretransplant stratified evaluation of risk of rejection, only kidney transplant recipients at high risk to develop CMV infection or disease, i.e., negative recipients of positive organ donors, patients receiving induction therapy with thymoglobulin and patients treated for acute rejection undergo preemptive strategy. Using this strategy, our currently overall incidence of CMV infection or disease is currently 25%. This incidence is higher among recipients who received thymoglobulin induction, tacrolimus and mycophenolate maintenance combination or treatment for acute rejection with either high dose of corticosteroids or thymoglobulin.

Because none of the kidney transplant recipients at our institution receive any prophylaxis for CMV infection and because immunosuppressive regimens are selected according to immunological rejection risk, this is the ideal population to investigate the natural history of CMV infection and disease using more recent, sensitive and specific molecular tolls.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent.
2. Male/female patients at least 18 years old who will be followed at our outpatient clinic for at least one year.
3. Recipients of first or repeat kidney transplants from living or deceased donors.

Exclusion Criteria:

1. Recipients of any combined transplant (kidney/pancreas, kidney liver).
2. Unlikely to comply with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All male and female de novo kidney transplant recipients
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Incidence of cytomegalovirus(CMV)infection and disease among renal transplant recipients receiving preemptive therapy. | 3 months
  There is still a debate regarding the superiority strategy with valganciclovir over the preemptive approach. Furthermore, this costly therapy or any other CMV prophylaxis is currently not reimbursed by our unified public health system. Therefore our strategy has been to use preemptive therapy.

SECONDARY OUTCOMES:
Change from baseline clinical and epidemiological aspects of CMV infection in this kidney transplant population. | 3 months
  Within each of these strategies, significant variation in clinical practice exists, including type of cellular or molecular diagnostics, antiviral therapies, monitoring and criteria for stopping treatment.We estimate that approximately 200 patients will be enrolled for this research. For this assessment we use monitoring for CMV replication:
  Samples will be collected every week for up to 3 months for determination of antigenemia and viral load. Investigators will be blinded to the results of the PCR analyses, unless unblinding is clinically indicated.
  Antigenemia test: Method: Antigen pp65 by indirect immunofluorescence. Reference: Zero Positive Cells /200.000 cells.
  Viral load test: Method: Real Time PCR - TaqMan Result: < 50 copies/mL Log: < 1.70 Detection Limit: 50 copies/mL Observations: Viral loads above 100 copies/mL should be considered active replication. Range of 50 to 109 copies/ml.
Incidence of the CMV viral load kinetics using a PCR-based assay among renal transplant recipients. | 3 months
  Questions include: (a) when after transplant is CMV viral load first detected; (b) how rapidly does viral load increase over time; and (c) what percent of patients with a detectable CMV viral load will develop a detectable CMV antigen.
The ideal time to start preemptive anti-CMV therapy. | 3 months
  Starting preemptive anti-CMV therapy based on viral load data. A question to consider is whether an absolute CMV viral load or a rate of change in the CMV.
Baseline factors that can predict those patients at risk for developing a CMV viral load parameter that correlates with development of a detectable CMV antigen. | 3 months
  Sorolical status CMV
Risk factors associated with prolonged treatment and recurrence of CMV infection or disease. | 3 months
  * Patients who have the serological status negative for cmv and received a kidney transplant from a donor with positive serology
  * Patients who underwent treatment for acute rejection
  * Patients who used thymoglobulin (induction and /or treatment of acute rejection)

CONTACTS AND LOCATIONS:
Overall Officials: Helio T Silva-Junior, MD, Principal Investigator — Hospital do Rim e Hipertensao
Locations (1):
- Hospital do Rim e Hipertensao, São Paulo, São Paulo, Brazil